CLINICAL TRIAL: NCT06852053
Title: Application to Predict Neonatal Apnea With Bradycardia (APNeA Study)
Brief Title: Application to Predict Neonatal Apnea With Bradycardia
Acronym: APNeA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Colm Travers, Associate Professor of Pediatrics, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 300008477; UAB (Other: UAB)
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-10

CONDITIONS: Apnea Neonatal; Bradycardia Neonatal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Virbrotactile stimulation (Experimental): Four hours of vibrotactile stimulation via a closed loop device if an apnea or bradycardia episode is predicted or detected.
  Interventions: Device: Closed-loop Vibro-Tactile Stimulator
- Control (Sham Comparator): Four hours of no vibrotactile stimulation via the closed loop device if an apnea or bradycardia episode is predicted or detected.
  Interventions: Device: Control

INTERVENTIONS:
Device: Closed-loop Vibro-Tactile Stimulator — Vibro-Tactile stimulation when bradycardia is predicted or predicted.
  Arms: Virbrotactile stimulation
Device: Control — Sham closed-loop vibrotactile stimulator
  Arms: Control

SUMMARY:
This purpose of this study is to reduce or stop apneas and bradycardias in pre-term infants, before they occur using gentle stimulation.

DETAILED DESCRIPTION:
This will be a randomized cross-over trial that will use additional ECG leads connected to a novel device and laptop to determine the accuracy and efficacy of an algorithm to predict, detect, and interrupt episodes of bradycardia for two 4-hour periods. There will be a 4-hour period without vibro-tactile stimulation and a 4-hour period with vibro-tactile stimulation when episodes are predicted or detected.

ELIGIBILITY:
Inclusion Criteria:

* Documented episodes of apnea with bradycardia over the previous 24 hours.
* Off ventilatory support/NCPAP for > 48 hours prior to study entry
* Gestational age < 32 0/7 weeks' gestation at birth
* Parents/legal guardians have provided consent for enrollment

Exclusion Criteria:

* a major malformation or a neuromuscular condition that affects respiration or causes apnea, or terminal illness or decision to withhold or limit support.

Ages: 22 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Bradycardia <100 beats per minute ≥ 10 seconds | 4-hours on either intervention.
  The frequency of episodes of bradycardia (heart rate less than 100 of ≥ 10 seconds) in either study arm during the study period.

SECONDARY OUTCOMES:
Bradycardia <60 beats per minute ≥ 5 seconds | 4 hours in either intervention.
  The frequency of episodes of bradycardia (heart rate <60 beats per minute ≥ 5 seconds) in either study arm during the study period.
Bradycardia <60 beats per minute ≥ 10 seconds | 4 hours on either intervention.
  The frequency of episodes of bradycardia (heart rate <60 beats per minute ≥ 10 seconds) in either study arm during the study period.
Bradycardia <80 beats per minute ≥ 5 seconds | 4 hours on either intervention.
  The frequency of episodes of bradycardia (heart rate <80 beats per minute ≥ 5 seconds) in either study arm during the study period.
Bradycardia <80 beats per minute ≥ 10 seconds | 4 hours on either intervention.
  The frequency of episodes of bradycardia (heart rate <80 beats per minute ≥ 10 seconds) in either study arm during the study period.
Proportion of time with Bradycardia < 100 beats per minute | 4 hours on either intervention.
  The total proportion of time with bradycardia during the study period on either intervention with a heartrate of <100 beats per minute.
Hypoxemia <85% for ≥ 5 seconds | 4 hours on either intervention.
  The frequency of episodes of hypoxemia (oxygen saturations <85% for ≥ 5 seconds) in either study arm during the study period.
Hypoxemia <85% for ≥ 10 seconds | 4 hours on either intervention.
  The frequency of episodes of hypoxemia (oxygen saturations <85% for ≥ 10 seconds) in either study arm during the study period.
Hypoxemia <90% for ≥ 5 seconds | 4 hours on either intervention.
  The frequency of episodes of hypoxemia (oxygen saturations <90% for ≥ 5 seconds) in either study arm during the study period.
Hypoxemia <90% for ≥ 10 seconds | 4 hours on either intervention.
  The frequency of episodes of hypoxemia (oxygen saturations <90% for ≥ 10 seconds) in either study arm during the study period.
Hypoxemia <80% for ≥ 5 seconds | 4 hours on either intervention.
  The frequency of episodes of hypoxemia (oxygen saturations <80% for ≥ 5 seconds) in either study arm during the study period.
Hypoxemia <80% for ≥ 10 seconds | 4 hours on either intervention.
  The frequency of episodes of hypoxemia (oxygen saturations <80% for ≥ 10 seconds) in either study arm during the study period.
Proportion of time with hypoxemia < 90% | 4 hours on either intervention.
  The total proportion of time with oxygen saturations <90% during the study period on either intervention.
Bradycardia prediction time | 4 hours on either intervention.
  The number of seconds ahead of routine patient monitors at which the device algorithm predicted bradycardia in either group.
Bradycardia prediction accuracy | 4 hours on sham control.
  The area under the curve for the true prediction rate over the false alarm rate in the control group.
Proportion of time with hypoxemia < 85% | 4 hours on either intervention.
  The total proportion of time with oxygen saturations <85% during the study period on either intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Colm P. Travers Associate Professor of Pediatrics, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be made available upon publication through a data use agreement to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal. Proposals should be submitted to cptravers@uabmc.edu.
Supporting Information: Study Protocol, SAP